CLINICAL TRIAL: NCT06469606
Title: A Cohort Study on feMale Patients' mammogRaphic texturE featureS: the COMPRESS Trial
Brief Title: Study on Female Patients' Mammographic Texture Features
Acronym: COMPRESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Kuopio University Hospital (Other); University of Eastern Finland (Other); University of Turku (Other); University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: R23077
Record Dates: First submitted 2024-05-30; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Artificial Intelligence; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant diagnosed with breast cancer (Experimental): Participants diagnosed with breast cancer who will undergo a mastectomy operation
  Interventions: Device: AI tool
- Participant not diagnosed with breast cancer (Experimental): Participants who will undergo a mastectomy operation for a non-breast cancer related clinical indication
  Interventions: Device: AI tool

INTERVENTIONS:
Device: AI tool — Both the arms will undergo the use of "AI tool" developed in the group. The tool will be trained to detect outcomes.

SUMMARY:
Mammography is the most common method for breast imaging, and it provides information for model building and analysis. Radiomics applied to mammography has the potential to revolutionize clinical decision-making by providing valuable insights into risk assessment and disease detection. Despite this, the influence of imaging parameters and clinical and biological factors on radiological texture features remains poorly understood. There is a pressing need to overcome the obstacle of system-inherent effects on mammographic images to facilitate the translation of radiological texture features into routine clinical practice by enabling reliable and robust AI-based or AI-aided decision-making. Furthermore, understanding the relationship between imaging parameters, textural features, and clinical and biological information supports the clinical use of AI. The objective of this study is to evaluate AI methods for clinical practice and to study how it relates to clinical factors and biological features.

ELIGIBILITY:
Inclusion Criteria:

* Candidate is a biological female aged 18 years or above;
* Candidate is willing and able to give informed consent and gives their written consent for the participation in the study;
* There is a clinical indication for a uni- or bilateral mastectomy

Exclusion Criteria:

* Candidate lacks the capacity to provide informed consent;
* Candidate has breast implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-17 (Estimated); Primary Completion 2035-12-15 (Estimated); Study Completion 2038-12-15 (Estimated)

PRIMARY OUTCOMES:
Mammographic texture features | Through study completion, an average of 5 year
  Aim: to evaluate how imaging parameters affect the mammographic texture features

SECONDARY OUTCOMES:
Biological features | through study completion, an average of 10 year
  Aim: To evaluate whether there is an interplay between mammographic texture feature parameters and pathological and biological features (e.g., breast cancer biomarkers)

IPD SHARING:
Plan to Share IPD: No